CLINICAL TRIAL: NCT04770168
Title: Harry Potter as a Novel Educational Paradigm to Improve Mental Wellness in Children: A Prospective Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Mark Sinyor, Associate Scientist/Psychiatrist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2200
Record Dates: First submitted 2021-02-12; First posted 2021-02-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Suicidal Ideation; Suicidal and Self-injurious Behavior; Suicide Attempt
Keywords: Suicidal ideation; Suicide attempts; Self-harm; Mental health literacy curriculum; School-based intervention; Cognitive behavioral therapy
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: This study employs a stepped wedge research design, allowing for both groups to receive the same cognitive behavioural therapy curriculum but during different time periods. Half the classes will receive the curriculum during the first half of the academic year and the rest of the classes will receive the curriculum during the second half of the academic year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT Curriculum - First Cohort (Experimental): Students will receive the 3-month cognitive behavioral therapy curriculum in the first half of the academic year.
  Interventions: Behavioral: Cognitive Behavioral Therapy Curriculum
- CBT Curriculum - Second Cohort (Waitlist Controls) (Experimental): Students will receive the current school board curriculum as usual for the first half of the academic year, serving as wait-list controls. Since this is a stepped wedge trial, the winter cohort will receive the identical intervention as the fall cohort in the second half of academic year.
  Interventions: Behavioral: Cognitive Behavioral Therapy Curriculum

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy Curriculum — The 3-month Harry Potter curriculum is delivered by trained teachers and includes lessons on a) risk factors that can contribute to emotional distress, b) how depression and anxiety manifest and how to access support/treatment, c) cognitive distortions, how they differ from rational thoughts and basic cognitive restructuring techniques, d) crisis planning including personalized "stressbusters" and "hope kits", and e) how to be resilient.

SUMMARY:
School-based mental health literacy interventions have been shown to reduce and/or prevent suicidal ideation and attempts. Most programs to date include an adapted version of Cognitive Behavioural Therapy (CBT) - the gold standard treatment for youth and adult mood and anxiety disorders. CBT teaches youth about the relationship between their thoughts, feelings, and behaviours, and provides strategies for managing distress. However, there is no established standard mental health literacy curriculum in Ontario. The investigators developed a school-based mental health literacy program that uses the third book in the Harry Potter series ('Harry Potter and the Prisoner of Azkaban') to teach students how to cope with distress through CBT skills. This study will determine whether the Harry Potter-based mental health literacy curriculum diminishes suicidality in students. The study will also determine whether the curriculum decreases depression and anxiety symptoms and improves well-being.

The 3-month intervention is a manual-based curriculum which teaches CBT skills in English class. The website includes video and text-based onboarding to train teachers on all the lessons. Youth complete online exercises for each unit and teachers follow a manual with checklists to preserve high fidelity and standardization of core learning.

Participating classes will be randomized in 1:1 fashion to receive the curriculum in the fall (~Oct-Dec) or the winter (~Feb-Apr). The study will use a stepped-wedge design to introduce the curriculum to classes sequentially testing whether students who receive it in fall will improve at mid-year and those in winter will catch up by year-end. The winter group is included as a "maturational" control to account for changes over the school year that are independent of the intervention and so that order effects of curriculum delivery can be tested. For this design, questionnaires will be administered four times throughout the school year (once before and after each semester), and once more the following year to measure duration of response. At each timepoint, subjects will complete validated questionnaires about suicide attempts and self-harm, anxiety, depression, well-being, and health services usage. Students may also choose to participate in focus groups to collect qualitative data on their experience with the curriculum. With additional consent (Ontario youth only), we will also collect aggregate lists of the Ontario Health Insurance Plan (OHIP) numbers for participating students. These will be provided to the Institute of Clinical Evaluative Sciences (ICES) who will identify sex, age and pre-existing healthcare utilization matched controls from regions that do not adopt the curriculum.

DETAILED DESCRIPTION:
Emerging evidence demonstrates that mental health literacy is a critical avenue for primary prevention of mental disorders as it increases awareness and recognition, decreases stigma, and encourages help-seeking. The largest mental health literacy study was conducted in Scandinavia and found that the combination of two lectures, three hours of role-play and an informational booklet reduced suicidal ideation and attempts after one year by approximately half in a cohort of more than 2,000 teenagers. The mental health literacy curriculum was the only intervention that was significantly better than a control group. The intervention has been piloted in more than 2,000 students in Ontario. The intervention is a 'literature study' taught over approximately 3 months in which a class reads the book and learns how distress and depression can manifest. The investigators have conducted two studies - a simple before and after design with 78 participants and a controlled trial with 200 participants who received the intervention and 230 wait list controls. Both indicated an intervention effect on suicide scores as well as improvements on a scale of symptoms of borderline personality disorder (e.g. emotional dysregulation), and depression and anxiety scores). These early findings suggest that this intervention may be a unique way of preventing suicidal ideation and attempts, and improving the mental health of youth across Canada and beyond.

The primary objective of the study is to determine whether the Harry Potter-based cognitive behavioural therapy curriculum diminishes suicidality (ideation and attempts) in students who receive it.

The primary hypothesis is that students receiving the curriculum will have a clinically and statistically significant reduction in rates (≥50%) on a composite measure of a) self-reported suicidal ideation, and b) self-reported suicide attempts.

Furthermore, the secondary objectives for the study are:

1. To determine whether the Harry Potter-based cognitive behavioural therapy curriculum decreases depression and anxiety symptoms and improves wellbeing immediately following the curriculum and approximately 6 months later.
2. To determine student and teacher satisfaction with the Harry Potter-based cognitive behavioural therapy curriculum
3. To create a website which achieves sufficient youth and teacher acceptability and 'youth friendliness' for widespread implementation

The secondary hypotheses are as follows:

1. Students receiving the curriculum will have a clinically and statistically significant reduction (≥50%) in their presentation to emergency services for self-harm/suicide attempts according to Ontario health administrative data (held in the Institute for Clinical Evaluative Services (ICES) repository). This is only applicable to research participants in Ontario.
2. Students receiving the curriculum will have clinically meaningful, significantly lower scores (≥25%) on validated instruments for youth depression and anxiety (the Revised Children's Anxiety and Depression Scale - RCADS), and wellbeing (the Life Problems Inventory - LPI) immediately after receiving it. Moreover, students will report a significant improvement (≥25%) on the Coping Scale for Children and Youth (CSCY) questionnaire.
3. Students in the first cohort (students who receive the curriculum in the fall semester) will have clinically meaningful, significantly lower scores (≥25%) on validated instruments for youth depression and anxiety (the Revised Children's Anxiety and Depression Scale - RCADS) and wellbeing (the Life Problems Inventory - LPI; Coping Scale for Children and Youth - CSCY) than the second cohort (students who receive the curriculum in the winter semester) at the mid-year point, but the two groups will not differ statistically at year end (i.e. the second cohort will catch up to the first).
4. There will be no significant difference between mid-year and year-end measures for the first cohort (i.e., gains will persist at approximately 6 months).
5. Student and teacher scores will both be high (mean ≥6 on 7-point Likert scales) on satisfaction questionnaires asking the degree to which they think they/their students benefited from the intervention, enjoyed the intervention, and would recommend it to others.
6. Student focus group data will reflect that students have experienced a qualitative improvement in wellbeing, knowledge of mental disorders and resilience following the curriculum.
7. Teacher interview data will reflect that teachers found the curriculum easy to implement and useful for imparting both mental health and general literacy to their students.
8. Students and teachers receiving the curriculum will achieve a mean score of ≥4 per question on a 5-point Likert-based questionnaire assessing acceptability and satisfaction as well as positive qualitative feedback.

ELIGIBILITY:
Inclusion Criteria:

* Only schools with Grade 7 and 8 classrooms (if requested, we may allow high school teachers/students in Grade 9 - 12 to participate as well)
* Participants must be able to speak and read fluent English
* Participants must be willing to complete demographic and clinical self-report questionnaires on anxiety, depression, and general well-being before the intervention and at each timepoint.

Exclusion Criteria:

-

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3204 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Composite of Self-Reported Suicidal Ideation and Attempts | Approximately 1-year period of study
  Composite includes self-reported suicidal ideation and self-reported suicide attempts, assessed by questions in the Life Problems Inventory (LPI).

SECONDARY OUTCOMES:
Presentation of Self-harm and Suicide Attempts | 1-year period of study
  Presentations to emergency services for self-harm/suicide attempts according to Ontario health administrative data (held in the Institute for Clinical Evaluative Services (ICES) repository). This is only applicable to research participants in Ontario.
Revised Children's Anxiety and Depression Scale | Approximately 1-year period of study
  Assesses youth depression and anxiety. Scale consists of 6 subscales, including Social Phobia (minimum score = 0, maximum score = 27), Panic Disorder (minimum score = 0, maximum score = 27), Major Depression (minimum score = 0, maximum score = 30), Separation Anxiety (minimum score = 0, maximum score = 21), Generalized Anxiety Disorder (minimum score = 0, maximum score = 18), and Obsessive-Compulsive (minimum score = 0, maximum score = 18). Higher scores indicate worse outcome.
Life Problems Inventory Questionnaire | Approximately 1-year period of study
  Assesses wellbeing and features borderline personality disorder. Minimum total score = 60. Maximum total score = 300. Higher scores indicate greater dysfunction and worse outcome. Subscales include confusion about self (minimum score = 15, maximum score = 75), impulsivity (minimum score = 15, maximum score = 75), emotional dysregulation (minimum score = 15, maximum score = 75), and interpersonal chaos (minimum score = 15, maximum score = 75).
Coping Scale for Children and Youth Questionnaire | Approximately 1-year period of study
  Assesses coping behaviours. Subscales include assistance seeking, cognitive-behavioural problem solving, cognitive avoidance, and behavioural avoidance. Higher scores indicate greater use of that coping dimension.
Student Satisfaction Questionnaire and Focus Group | Approximately 1-year period of study
  Composite of responses from self-report questionnaires and focus groups which assesses the degree to which students benefitted from the intervention, enjoyed the intervention, and would recommend to others. Higher scores indicate greater satisfaction.
Teacher Satisfaction Questionnaire and Focus Group | Approximately 1-year period of study
  Composite of responses from self-report questionnaires and focus groups which assesses the degree to which teachers think that their students benefitted from the intervention, enjoyed the intervention, and would recommend to others. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- See also: Website for the MyOwl website which contains all the lesson plans and student activities for the curriculum. — http://www.myowl.org